CLINICAL TRIAL: NCT04271878
Title: Hypercapnia and Orthostatic Tolerance in Postural Orthostatic Tachycardia Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REB20-0135
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Postural Tachycardia Syndrome; Orthostatic Intolerance
Keywords: postural tachycardia; autonomic; orthostatic intolerance; dysautonomia
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance; Autonomic Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: All participants must have been diagnosed with POTS, they will all complete up to 6 head-up tilt tests (HUTTs) on a single day. They will all receive the following interventions:
  1. Normal not coached breathing and room air
  2. Normal not coached breathing with ETCO2 clamped at baseline levels - The baseline CO2 levels will be defined from the mean end-tidal CO2 (ETCO2) measured through the mask over the last 5 min of the first baseline phase (ETCO2 normal values range between 35mmHg and 45mmHg).
  3. Normal not coached breathing with mild ETCO2 levels (45mmHg)
  4. Normal not coached breathing with high ETCO2 levels (55mmHg)
  5. Fast breathing and resultant low ETCO2 levels (target ETCO2 19-24mmHg);
  6. Fast breathing and ETCO2 clamped at baseline levels
Masking Description: All participants will be fitted with a face mask connected to a tube supplied with gas from the RespirAct™ system. The participants will not be informed about the concentration of gases during the tilt tests. After the study completion they will be informed about the order of interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Other): All participants will receive the same interventions
  Interventions: Other: RespirAct™ system (Thornhill Research Inc., Toronto, Canada)

INTERVENTIONS:
Other: RespirAct™ system (Thornhill Research Inc., Toronto, Canada) — 1. HUTT with Normal Breathing in Room Air (No gas interventions will be applied)
  2. HUTT with Normal Breathing and ETCO2 clamped at baseline levels
  3. HUTT with Normal Breathing and Mild Hypercapnia (the ETCO2 will be clamped at 45mmHg )
  4. HUTT with Normal Breathing and High Hypercapnia (the ETCO2 will be clamped at 55mmHg)
  5. HUTT with Fast, Deep Breathing and resultant Hypocapnia Participant will be coached to breath around 15 breath per min.No gas interventions will be applied
  6. HUTT with Fast, Deep Breathing and ETCO2 clamped at baseline levels. Participant will be coached to breath around 15 breath per min, with ETCO2 clamped to baseline levels.

SUMMARY:
The mechanism behind postural orthostatic tachycardia syndrome (POTS) involves many causes including a sympathetic nervous system problem. Blood gases, like carbon dioxide (CO2), have an important effect on sympathetic activation.

The purpose of this research study is to determine if higher CO2 levels have any effect in lowering heart rate and reducing POTS symptoms when upright/standing. The investigators are also searching for the ideal CO2 concentration to achieve the most effective response

DETAILED DESCRIPTION:
The effects of hypercapnia on cerebral blood flow velocity and arterial blood pressure in healthy subjects lead to an increase in orthostatic tolerance, peak HR and time to peak HR compared with normocapnic orthostatism. The CO2 effects on heart rate and orthostatic tolerance were observed in a small group of POTS patients with orthostatic hypocapnia, after supplying CO2 to correct hypocapnia. It is unclear, however, whether this intervention will also work for the broader POTS population. This might constitute an attractive option of therapy for POTS patients.

The investigator's hypothesis is that increasing end-tidal CO2 (ETCO2) will reduce orthostatic tachycardia and orthostatic symptoms in patients with POTS. The secondary hypothesis is that blood pressure will be better maintained during increased ETCO2 via improved cardiac output.

INTERVENTION The RespirAct™ system (Thornhill Research Inc., Toronto, Canada) is a computer-controlled gas blender providing CO2, O2 and nitrogen for a subject to inhale while breathing for the purpose of controlling the concentrations of the respective blood gases. The RespirAct™ records inspired and exhaled gas concentrations, which can be recalled, analyzed and graphed. Data is collected breath-by-breath including end-tidal O2 and CO2, the length of inspiration and expiration for the breath, the respiration rate and the tidal volume per breath. The system has been Health Canada approved and utilized in several publications in healthy individuals and clinical populations. Subjects will be fitted with a face mask which will be connected to a tube supplied with gas from RespirAct™ system

Primary Analysis The primary analysis will compare the magnitude of ΔHR from supine to HUTT during hypercapnia compared to HUTT with no intervention (HUTT 3 and 4 vs 1). The comparison will use a paired t-test (or a Wilcoxon Signed-Rank test if the data are non-normally distributed).

Secondary Analysis The secondary analysis will compare the VOSS Symptom Rating at the end of each 8 min HUTT, comparing each HUTT run.

Sample Size Calculation Since this is a pilot study, there are few preliminary data about the effect of hypercapnia on orthostatic symptoms in POTS adults. A clinically meaningful reduction in orthostatic tachycardia of 10 bpm would be clinically significant. It is estimated a standard deviation of about 15 bpm for our sample. With the aforementioned assumptions for a paired test of continuous data and a 0.05 two-sided significance level, a sample size of 20 POTS patients would allow for 80% power to detect this difference. To account for study withdrawal and dropout the investigators intend to enroll 26 POTS patients in total

Adverse Event (or Unanticipated Problem) Reporting Any adverse events of a serious nature will be reviewed immediately with the principal investigator. Serious adverse events will be reported in writing to the CHREB within 10 days of the PI's notification of the event. All study adverse events will be summarized once a year, during the annual review reporting, for the CHREB. The research coordinator will be responsible for tracking adverse events in this study.

The adverse event will be described with the following information: description of the event, outcome of the event, how long it lasted, whether the event required treatment or intervention, and the outcome.

The definition of events is as follows:

Mild - transient and mild in nature, with no treatment necessary. Moderate - some intervention and treatment necessary, but the participant completely recovers. Severe - an event that results in hospitalization, disability, death or is life-threatening.

Data & Safety Monitor There will be no external Data & Safety monitor for this study.

PRIVACY and CONFIDENTIALITY ISSUES

Protected Health Information will be used in this study. The investigators will comply with the patient privacy guidelines of the University of Calgary and applicable provincial and federal rules.

The research team is comprised of experienced research nurses and research assistants who are aware of the importance of confidentiality of health information. Paper research records will be stored in a locked office. Digital records will be stored on password-protected University of Calgary computers/servers and in the University of Calgary Clinical Research Unit REDCap Database.

Every effort will be made to publish and present the data from this study. At no time will any participant be identified in any such publication

Information about participants will be handled as confidentially as possible, but there is always the potential for an unintended breach of privacy.

Data Management Plan:

* All data will be stored under an assigned participant code for data storage and a master list linking the code to the participant name and other identifiers will be kept on the encrypted restricted access drive at the University of Calgary.
* All data collected before, during, and after the study, including identifiable data, will always be kept on password protected computers on an encrypted restricted access drive at the University of Calgary or in the case of paper records, locked in a secure file cabinet in a locked room. Only the researchers will have access to these.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of Postural Tachycardia Syndrome (POTS)
* Age 18-60 years
* Male and Female
* Non - smokers.
* Able and willing to provide informed consent.
* Ability to travel to Libin Cardiovascular Institute of Alberta Autonomic Testing Lab at the University of Calgary, Calgary, AB.

Exclusion Criteria:

* Overt cause for postural tachycardia, i.e., acute dehydration
* Participants with somatization or severe anxiety symptoms will be excluded
* Pregnant
* Inability to tolerate mask for the duration of the study
* Subjects who require portable oxygen at rest or with exercise
* Subjects with chronic heart failure or severe pulmonary disease who are unable to climb one flight of stairs due to shortness of breath.
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Heart Rate (HR) variation | difference between HR from supine to peak HR during tilt test for each intervention (mean value HR between the 8th and 9th minute of supine; peak parameters, during HUTT, mean value during the first min and between the 3rd and 8th min)
  Magnitude of ΔHR

SECONDARY OUTCOMES:
Cerebral blood flow velocity (CBFv) variation | difference between CBFv from supine to peak during tilt test for each intervention (mean value CBFv between the 8th and 9th min of supine; peak parameters, during HUTT, mean value CBFv during the first min and between the 3rd and 8th min)
  Magnitude of ΔCBFv
VOSS symptom score | VOSS will be accessed at the 8th minute of each HUTT, comparing the intensity of symptoms in each intervention
  Vanderbilt Orthostatic Symptoms Score (VOSS) - patients will rate the severity of 9 symptoms on a scale of 0 to 10 (0 reflects absence of symptoms). The sum of the scores at each time point is used as a measure of symptom burden (lower score reflects reduced symptom burden). The 9 symptoms are mental clouding, blurred vision, shortness of breath, rapid heartbeat, tremulousness, chest discomfort, headache, lightheadedness, and nausea.

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD, MSCI, Principal Investigator — University of Calgary, Cardiac Science
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Del Pozzi AT, Schwartz CE, Tewari D, Medow MS, Stewart JM. Reduced cerebral blood flow with orthostasis precedes hypocapnic hyperpnea, sympathetic activation, and postural tachycardia syndrome. Hypertension. 2014 Jun;63(6):1302-8. doi: 10.1161/HYPERTENSIONAHA.113.02824. Epub 2014 Apr 7. PMID 24711524
- [Background] Ocon AJ, Medow MS, Taneja I, Clarke D, Stewart JM. Decreased upright cerebral blood flow and cerebral autoregulation in normocapnic postural tachycardia syndrome. Am J Physiol Heart Circ Physiol. 2009 Aug;297(2):H664-73. doi: 10.1152/ajpheart.00138.2009. Epub 2009 Jun 5. PMID 19502561
- [Background] Taneja I, Medow MS, Clarke DA, Ocon AJ, Stewart JM. Baroreceptor unloading in postural tachycardia syndrome augments peripheral chemoreceptor sensitivity and decreases central chemoreceptor sensitivity. Am J Physiol Heart Circ Physiol. 2011 Jul;301(1):H173-9. doi: 10.1152/ajpheart.01211.2010. Epub 2011 May 2. PMID 21536847
- [Background] Stewart JM, Pianosi P, Shaban MA, Terilli C, Svistunova M, Visintainer P, Medow MS. Postural Hyperventilation as a Cause of Postural Tachycardia Syndrome: Increased Systemic Vascular Resistance and Decreased Cardiac Output When Upright in All Postural Tachycardia Syndrome Variants. J Am Heart Assoc. 2018 Jun 30;7(13):e008854. doi: 10.1161/JAHA.118.008854. PMID 29960989
- [Result] Novak P. Hypocapnic cerebral hypoperfusion: A biomarker of orthostatic intolerance. PLoS One. 2018 Sep 26;13(9):e0204419. doi: 10.1371/journal.pone.0204419. eCollection 2018. PMID 30256820